CLINICAL TRIAL: NCT00672503
Title: "Decreasing Catheter-Associated Urinary Tract Infections in the Pediatric Intensive Care Unit
Brief Title: Decreasing Catheter-Associated Urinary Tract Infections in the Pediatric Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Tangela Welch, RN, PICU Clinical Research Coordinator, Children's Mercy Hospital Kansas City
Other Study IDs: 08 04-065E
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Urinary Tract Infections
Keywords: indwelling urinary catheters; urinary tract infections; foley-catheter related infections; hospital acquired CA-UTI
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Patients who acquired a CA-UTI in the PICU between 2004-2007.
- 2: Patients who did not acquire a CA-UTI while hospitalized in the PICU but had an indwelling urinary catheter between 2004-2007.
- A: Nurses currently employed in the PICU at Children's Mercy Hospital.
- a: Root Cause Analysis on all patients who acquired a CA-UTI during 2009.

SUMMARY:
The purpose of this study is to identify risk factors associated with indwelling urinary catheters, as well as to assess the nurses' knowledge and adherence to hospital policies. The study will also include a very extensive literature search in an attempt to create a national standard or guideline.

ELIGIBILITY:
Inclusion Criteria:

1. Medical records of 67 patients 0 to 17 years of age diagnosed with a catheter associated urinary tract infection (defined by CDC) acquired during a PICU hospitalization.
2. Medical records of 67 patients 0 to 17 years of age who had an indwelling urinary catheter during a PICU hospitalization without a catheter associated urinary tract infection.
3. Nurses employed at Children's Mercy Hospital in the PICU.
4. Patient's who acquired a CA-UTI during 2009 and was adjudicated by infection control.

Exclusion Criteria:

Patients

1. Patients with community acquired urinary tract infections
2. Patients 18 years and older cared for in the PICU.
3. Patients with catheter associated urinary tract infections hospitalized outside the PICU at Children's Mercy Hospital.
4. Patients with UTI not related to catheterization

Nurses

1. Nurses floated to the PICU who are not permanent staff members (ICN nurse, float pool staff, travelers)
2. Nurses on the research team

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 1. Patients who acquired a CA-UTI while hospitalized in the PICU between 2004-2007.
  2. Patients who had an indwelling urinary catheter while hospitalized in the PICU between 2004-2007 but did not acquire a CA-UTI.
  3. Nurses currently employed in the PICU at Children's Mercy Hospital.
  4. All Patient's who acquired a CA-UTI during 2009
Sampling Method: Non-Probability Sample
Enrollment: 321 (Actual)
Dates: Start 2008-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Identification of risk factors associated with indwelling urinary catheters. | 2004-2007

SECONDARY OUTCOMES:
Identification of nurses' knowledge of insertion, irrigation, care and maintenance of indwelling urinary catheters. | 2008

CONTACTS AND LOCATIONS:
Overall Officials: Tangela M Welch, ADN, BBA, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospitals and Clinics, Kansas City, Missouri, United States